CLINICAL TRIAL: NCT02459886
Title: A Phase 1 Randomized, Double-Blinded, Placebo-Controlled Single-Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB054 in Healthy Subjects and Subjects With Early Parkinson's Disease
Brief Title: Single-Ascending Dose Study of BIIB054 in Healthy Participants and Early Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 228HV101
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Parkinson's Disease; Healthy
Keywords: alpha synuclein; PD
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Single intravenous (IV) low dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo
- Cohort 2 (Experimental): Single IV ascending dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo
- Cohort 3 (Experimental): Single IV ascending dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo
- Cohort 4 (Experimental): Single IV ascending dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo
- Cohort 5 (Experimental): Single IV ascending dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo
- Cohort 6 (Experimental): Single IV ascending dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo
- Cohort 7 (Experimental): Single IV ascending dose infusion with staggered participant dosing
  Interventions: Drug: BIIB054; Drug: Placebo

INTERVENTIONS:
Drug: BIIB054 — IV infusion
Drug: Placebo — IV infusion

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of a range of single BIIB054 doses, administered as a single intravenous (IV) infusion, in healthy participants and participants with early Parkinson's disease (PD). Secondary objectives of the study are to assess the serum pharmacokinetics (PK) profile of BIIB054 after single-dose administration and to evaluate the immunogenicity of BIIB054 after single-dose administration.

DETAILED DESCRIPTION:
Only healthy participants will be enrolled in Cohorts 1 through 6. Only participants with early PD will be enrolled in Cohort 7

ELIGIBILITY:
Key Inclusion Criteria:

1. All women of childbearing potential and all men must practice effective contraception during the study and for 6 months after their last dose of study treatment.
2. Must have a body mass index from 19 to 32 kg/m2, inclusive.
3. Must be in good health as determined by the Investigator, based on medical history, physical examination, and 12-lead ECG.

   For cohort 7 only:
4. Diagnosis of idiopathic PD

Key Exclusion Criteria:

1. History of cardiovascular disease.
2. Subject smokes more than 5 cigarettes or the equivalent in tobacco daily.
3. Surgery within 3 months prior to Day -1 (other than minor cosmetic surgery and minor dental surgery, as determined by the Investigator).
4. History or positive test result for hepatitis C, hepatitis B, or human immunodeficiency virus (HIV).
5. Female subjects who are pregnant, currently breastfeeding, or attempting to conceive during the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Adverse events/serious adverse events (AEs/SAEs), | 20 Weeks
  After a range of single BIIB054 doses administered as a single IV infusion in healthy participants and participants with early Parkinson's Disease, clinical laboratory test data, vital signs, neurological and physical examination findings, 12-lead electrocardiogram (ECG) data, and brain magnetic resonance imaging (MRI) findings will be used in the evaluation of AEs/SAEs.
Columbia Suicide Severity Rating Scale (C-SSRS) | 20 Weeks
  The Columbia Suicide Severity Rating Scale, or C-SSRS, is a suicidal ideation rating scale created by researchers at Columbia University to evaluate suicidality.
Montreal Cognitive Assessment (MoCA) | 20 Weeks
  The Montreal Cognitive Assessment MoCA is a brief cognitive screening tool for Mild Cognitive Impairment.

SECONDARY OUTCOMES:
Evaluate serum BIIB054 concentrations and PK parameters | 20 Weeks
  Area under the concentration-time curve (AUC) from time zero extrapolated to infinity (0-∞), AUC from time 0 to time of the last measurable concentration (AUC0-tlast), maximum concentration (Cmax), time to Cmax (Tmax), elimination half-life (t1/2), and clearance (Cl), will be used to assess the serum PK profile of BIIB054 after single-dose administration.
evaluation of anti-BIIB054 antibodies in serum | 20 Weeks
  evaluate the immunogenicity of BIIB054 after single-dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (9):
- United States (9):
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Hallandale, Florida
  - Research Site, Oviedo, Florida
  - Research Site, Evansville, Indiana
  - Research Site, Farmington Hills, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Dallas, Texas
  - Research Site, Spokane, Washington